CLINICAL TRIAL: NCT03790995
Title: Intermediate Term Functional Outcomes and Quality of Life in Patients With High Versus Low and Intermediate Risk Prostate Cancer Treated by Robot-assisted Laparoscopic Prostatectomy (RALP)
Brief Title: Functional Outcomes and QoL in Patients With High Versus Low and Intermediate Risk Prostate Cancer Treated by RARP
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Belgian Cancer Registry (Other)
Responsible Party: Principal Investigator, Wout Devlies, Principal Investigator, KU Leuven
Other Study IDs: Be-RALP functioning and QoL
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer; Quality of Life; Erectile Function; Urinary Function
Keywords: Prostate cancer; Robot assisted radical prostatectomy; RALP; RARP; High risk; Intermediate risk; Low risk; Urinary; Erectile; Quality of life; QoL; Post operation; functional outcomes; follow-up
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk prostate cancer: Patients with initial cT2c-3-4, cN +, Gleason score (GS) more than 7 or PSA > 20ng/mL were labelled as high-risk prostate cancer.
  Both groups received robot assisted laparoscopic prostatectomy. Matching across age (continuous), year of surgery (2009+2010, 2011, 2012, 2013, 2014, 2015+2016), nerve sparing (bilateral, unilateral or no nerve sparing) and centre size (continuous). 1:1 coarsened exact matching. Continuous variables are temporarily coarsened as followed: age (<55, 55-<65, 65-<75, 75+) and centre size (<50, 50-<100, 100+ cases/year).
  Interventions: Procedure: Robot assisted laparoscopic prostatectomy
- Low - intermediate risk prostate cancer: Initial PSA levels less or equal than 20 ng/mL with GS of 7 or less and cT1-2a-2b, 2 were labelled as low and intermediate risk prostate cancer and served as a control group.
  Both groups received robot assisted laparoscopic prostatectomy. Matching across age (continuous), year of surgery (2009+2010, 2011, 2012, 2013, 2014, 2015+2016), nerve sparing (bilateral, unilateral or no nerve sparing) and centre size (continuous). 1:1 coarsened exact matching. Continuous variables are temporarily coarsened as followed: age (<55, 55-<65, 65-<75, 75+) and centre size (<50, 50-<100, 100+ cases/year).
  Interventions: Procedure: Robot assisted laparoscopic prostatectomy

INTERVENTIONS:
Procedure: Robot assisted laparoscopic prostatectomy
  Other Names: +- postoperative treatments

SUMMARY:
The Be-RALP database is Belgian prospective multicenter database governed by the Belgian cancer registry. This database investigates the status after robot assisted laparoscopic prostatectomy (RALP) in prostate cancer patients. It was established by a collaboration between the Belgian association of Urology (BAU), the National Institute for Health and Disability Insurance (NIHDI) and the Belgian cancer registry.

Between 2009 and 2016, 9235 patients were included in this patient registry.

The studied outcomes covered quality of life measures as well as variables covering urinary and erectile function.

DETAILED DESCRIPTION:
The Be-RALP database is Belgian prospective multicenter database governed by the Belgian cancer registry. This was established by a collaboration between the Belgian association of Urology (BAU), the National Institute for Health and Disability Insurance (NIHDI) and the Belgian cancer registry.

Twenty-five centres, on average 90% of all Belgian robotic centres, collected prospective data of 9235 patients from October 2009 until February 2016. These data is collected by local data managers or physicians and was required to receive reimbursion from the NIHDI for the disposables used during robot surgery. After filling in the data by the local datamanagers, the data is centralised. In Brussels the data is protected and further used by data managers and statisticians. In this system in-and output of data is strictly separated. Patient data is encoded to ensure absolute privacy. Then the data is checked upon correctness by using random checks. Data is completed where necessary.

These parameters increase the quality of data handling and database.

The final database consists of baseline pre-, per- and postoperative data as well as four standardised follow-up registrations (on 1, 3, 12 and 24 months), with follow-up data still being collected. In each follow-up registration, functional parameters and quality of life are re-assessed together with postoperative treatment status and PSA.

The Be-RALP database collected patient details of 9235 patients treated by RARP between 2009 and 2016. Patients with macro metastasis and initial PSA values higher than 100 (probable undetected micro metastasis) were excluded for this study, as well as all pT0, patients with surgery after the closing date and patients with invalid survival data. Further exclusion of patients with missing values for nerve sparing, extend of nerve sparing and risk category resulted in a group of 8306 patients.

The selected outcomes covered in the database consist of quality of life measures (European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 global, physical, emotional and cognitive) as well as variables covering urinary (Incontinence Modular Questionnaire-Urinary Incontinence: ICIQ, EORTC QLQ-PR25 urinary symptoms, incontinence aid) and erectile function (International Index of Erectile Function: IIEF, EORTC QLQ-PR25 sexual activity and sexual functioning).

A 1:1 matching between high and low-intermediate prostate cancer will be performed. Afterwards, longitudinal mixed models will quantify the relation between the explanatory variables follow-up time, risk group (high vs. low-intermediate) and postoperative treatment (postoperative radiotherapy (RT) and/or androgen deprivation therapy (ADT): yes vs. no) and the outcomes erectile- and urinary function as well as Quality of Life. All analysis will be performed using the statistical analysis software (SAS system), version 9.3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer
* Eligible to undergo RALP
* RALP in one of the 25 participating centres

Exclusion Criteria:

* iPSA > 100
* Confirmed metastasis
* invalid survival data
* pT0
* Missing nerve sparing details
* Missing risk group

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from 90% of all Belgian robotic assisted radical prostatectomy centres between 2009 and 2016 with prostate cancer undergoing RALP. Patients reflect very well the Belgian prostate cancer patient population since 25 centres participated.
  NIHDI reimbursement criteria insured a high inclusion rate.
Sampling Method: Non-Probability Sample
Enrollment: 9235 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Global quality of life | Longitudinal modelling over 24 months
  EORTC C30 global quality of life, questionnaire
Emotional quality of life | Longitudinal modelling over 24 months
  EORTC C30 emotional quality of life, questionnaire
physical quality of life | Longitudinal modelling over 24 months
  EORTC C30 physical quality of life, questionnaire
Cognitive quality of life | Longitudinal modelling over 24 months
  EORTC C30 cognitive quality of life, questionnaire
Erectile function - IIEF 5 | Longitudinal modelling over 24 months
  International Index of Erectile Function (IIEF-5), questionnaire
Erectile function - sexual activity | Longitudinal modelling over 24 months
  EORTC PR25 sexual activity, questionnaire
Erectile function - sexual functioning | Longitudinal modelling over 24 months
  EORTC PR25 sexual functioning, questionnaire
Urinary function - Incontinence aid | Longitudinal modelling over 24 months
  EORTC PR25 incontinence aid, questionnaire
Urinary function - urinary symptoms | Longitudinal modelling over 24 months
  EORTC PR25 urinary symptoms, questionnaire
Urinary function - ICIQ | Longitudinal modelling over 24 months
  International Consultation on Incontinence Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joniau, Professor, Principal Investigator — Department of Urology, KU Leuven, Leuven Belgium
Locations (25):
- Belgium (25):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze-Lieve-Vrouwziekenhuis Aalst-Asse-Ninove, Aalst
  - GZA ziekenhuizen - Campus Sint-Augustinus, Antwerp
  - AZ Klina, Brasschaat
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - AZ Sint-Lucas, Bruges
  - CHU Saint-Pierre Bruxelles, Brussels
  - Institut Jules Bordet Bruxelles, Brussels
  - Hôpital Erasme Bruxelles, Brussels
  - CHIREC, Brussels
  - AZ Sint Blasius Dendermonde, Dendermonde
  - AZ Jan Palfijn Gent, Ghent
  - AZ Maria Middelares Gent, Ghent
  - AZ Sint-Lucas Gent, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Universitaire ziekenhuizen Leuven, Leuven
  - CHR de la Citadelle Liège, Liège
  - CHU Ambroise Paré Mons, Mons
  - AZ Damiaan, Ostend
  - AZ Delta-Heilig Hart Ziekenhuis Roeselare-Menen, Roeselare
  - Cliniques de l'Europe Bruxelles, Uccle
  - AZ Jan Portaels, Vilvoorde
  - Cliniques Universitaires de Mont-Godinne, Yvoir
  - AZ Sint-Elisabeth Zottegem, Zottegem

IPD SHARING:
Plan to Share IPD: No
After discussion with the board on the requested data, possibly aggregated data can be send to the requesting party.
  No individual patient data can be send due to privacy concerns and local legislations

REFERENCES:
- [Background] Albisinni S, Joniau S, Quackels T, De Coster G, Dekuyper P, Van Cleynenbreugel B, Van Damme N, Van Eycken E, Ameye F, Roumeguere T; Be-RALP Registry (Belgian Robotic-Assisted Laparoscopic Prostatectomy Registry). Current trends in patient enrollment for robotic-assisted laparoscopic prostatectomy in Belgium. Cancer. 2017 Nov 1;123(21):4139-4146. doi: 10.1002/cncr.30874. Epub 2017 Jul 25. PMID 28743170
- [Background] Tosco L, De Coster G, Roumeguere T, Everaerts W, Quackels T, Dekuyper P, Van Cleynenbreugel B, Van Damme N, Van Eycken E, Ameye F, Joniau S; Be RALP the Belgian RALP consortium. Development and External Validation of Nomograms To Predict Adverse Pathological Characteristics After Robotic Prostatectomy: Results of a Prospective, Multi-institutional, Nationwide series. Eur Urol Oncol. 2018 Sep;1(4):338-345. doi: 10.1016/j.euo.2018.04.008. Epub 2018 Jun 7. PMID 31100256